CLINICAL TRIAL: NCT07021027
Title: Feasibility Study of Whole Egg Consumption in Adults With Intermediate Age-related Macular Degeneration
Brief Title: Eggs and Age-related Macular Degeneration (EggsAMD) Study.
Acronym: EggsAMD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kathryn Starr (Other)
Responsible Party: Sponsor-Investigator, Kathryn Starr, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00112553
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Intermediate Age-Related Macular Degeneration
Keywords: Intermediate Age-Related Macular Degeneration; Older Adults; Eggs; vision

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Whole Egg - 4 (Experimental): Participants will be asked to consume 4 medium eggs per day for five months.
  Interventions: Drug: Whole Egg - 4
- Whole Egg - 2 (Active Comparator): Participants will be asked to consume 2 medium eggs per day for five months.
  Interventions: Drug: Whole Egg - 2

INTERVENTIONS:
Drug: Whole Egg - 4 — Participants will be asked to consume 4 medium Eggland's Best eggs per day for 5 months.
  Arms: Whole Egg - 4
Drug: Whole Egg - 2 — Participants will be asked to consume 2 medium Eggland's Best eggs per day for 5 months.
  Arms: Whole Egg - 2

SUMMARY:
Age-related macular degeneration (AMD) is the primary cause of vision loss in people over the age of 55. Currently, no cure is available for individuals suffering from AMD. The purpose of this pilot study is to evaluate the feasibility of implementing a 5-month egg intervention in adults with intermediate AMD. The objective of this research study is to evaluate the feasibility of a whole egg (2 or 4 per day) intervention in older adults with intermediate AMD. The secondary objective of this research is to determine descriptive statistics, change over time and estimate effect sizes for retinal sensitivity, and vision, cognition and physical function. By completing these research objectives, the researchers hope to gain preliminary evidence in support of a larger trial that will assess the impact of egg consumption on eye health in adults with AMD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with intermediate dry AMD as noted in their medical record (defined as having multiple medium drusen, at least one large druse (>125 μm or the approximate size of a vessel coming off the optic nerve), and/or non-center involving geographic atrophy) who are BCVA stable from prior exam within 6 months - defined by change of < 10 letters on EDTRS chart (BCVA within 10 letters within past 6 months)
* 55 years of age and older
* Willing to limit consumption of eggs for one month prior to beginning the study intervention
* Willing to follow diet protocol
* Body Mass Index (22.0 - 39.9 kg/m2)
* Access to refrigeration
* Access to reliable transportation

Exclusion Criteria:

* Presence of retinal pathology such as central geographic atrophy, hemorrhage or retinal fluid and other macular pathology other than AMD
* Presence of dense cataracts
* Presence of glaucoma
* Previous retinal laser or surgical therapy that has impacted the integrity of the retina
* Any other ocular condition requiring long-term therapy or surgery during the study period
* Participant has photographically significant corneal or media opacities in either eye that would preclude adequate ophthalmic imaging and functional testing
* Diagnosis of nystagmus that will interfere with testing
* Egg allergy
* Uncontrolled hyperlipidemia (cholesterol >240 mg/dL in the last 12 months, unless under active medication management to achieve <240 mg/dL)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adherence rate to consuming four whole eggs per day | From intervention start to the end of treatment at 5 months.
  Adherence Rate (%) = (Number of days with 4 whole eggs consumed / Total number of days in the observation period) x 100

SECONDARY OUTCOMES:
Vision function, as measured by percent reduced threshold (PRT) | Baseline and 5 months
  Mesopic microperimetry with eye tracking (MAIA) results will be reported as percent reduced threshold (PRT), defined as the percentage of abnormal retinal sensitivity thresholds below 25 dB.
Vision function, as measured by Average threshold (AT) | Baseline and 5 months
  Mesopic microperimetry with eye tracking (MAIA) results will be reported as average threshold (AT), defined as the average of retinal sensitivity values from all loci tested.
Vision function, as measured by Central macular thickness | Baseline and 5 months
  Central macular thickness will be measured by Optical Coherence Tomography (OCT)
Vision function, as measured by Best Corrected Visual Acuity (BCVA) | Baseline and 5 months
  BCVA will be assessed by reading a standard eye chart placed at a distance
Vision function, as measured by Low Luminance Visual Acuity (LL-BCVA) | Baseline and 5 months
  LL-BCVA will be assessed by reading a standard eye chart placed at a distance in low-light conditions
Vision function, as measured by Reading Acuity (MN Read) | Baseline and 5 months
  Participants will be asked to read a chart with various print sizes (MNREAD acuity charts)
Vision function, as measured by Contrast Sensitivity | Baseline and 5 months
  Participants will be asked to read letters (which will be colored in a range of gray) on an eye chart or iPad, placed at a distance.
Vision function, as measured by National Eye Institute Visual Functioning Questionnaire - 25 (VFQ-25) | Baseline and 5 months
  Participants will rate their vision on multiple activities of daily living based on their own opinion. The NEI VFQ-25 is scored by converting item responses to a 0-100 scale, averaging them into subscales, and calculating a composite score (excluding general health), with higher scores indicating better visual function.
Cognitive function, as measured by the Hopkins Verbal Learning Test | Baseline and 5 months
  The Hopkins Verbal Learning Test is scored by summing the number of correct words recalled across three learning trials (Total Recall), the number recalled after a delay (Delayed Recall), and the number of correctly identified words on a recognition task (Recognition Discrimination Index), with higher scores indicating better verbal learning and memory performance.
Physical Function, as measured by balance | Baseline and 5 months
  Will be asked to stand for 10 seconds with feet in 3 different positions (side-by-side, semi-tandem, tandem). The balance component of the SPPB is scored from 0 to 4 based on the ability to hold side-by-side, semi-tandem, and tandem stances for up to 10 seconds each, with higher scores indicating better balance.
Physical Function, as measured by 30-Second Chair Stand | Baseline and 5 months
  Number of full stands that can be completed in 30 seconds with arms folded across chest
Physical Function, as measured by 30-Second Arm curl | Baseline and 5 months
  Number of arm curls completed in 30 seconds.
Physical Function, as measured by 8-foot up and go | Baseline and 5 months
  Number of seconds required to get up from a seated position, walk 8 feet (2.44 m), turn, and return to seated position
Quality of Life, as measured by the 36-Item Short Form Health Survey (SF-36) | Baseline and 5 months
Dietary Intake | Baseline and 5 months
  3-day food record and recalls. Total calories (kcals) consumed are determined by averaging the intake of three days. A higher mean number indicates that more calories are consumed.
Satisfaction with study participation | From enrollment to the end of treatment at 5 months
  On a 1-5 Likert scale (1 = Very Dissatisfied, 5 = Very Satisfied), overall, how satisfied are you with your decision to participate in this study?
Satisfaction with egg consumption (Whole Egg - 2) | From intervention start to the end of treatment at 5 months.
  On a 1-5 Likert scale (1 = Very Dissatisfied, 5 = Very Satisfied), How satisfied were you with consuming two medium eggs per day for the duration of the study?
Satisfaction with egg consumption (Whole Egg - 4) | From intervention start to the end of treatment at 5 months.
  On a 1-5 Likert scale (1 = Very Dissatisfied, 5 = Very Satisfied), how satisfied were you with consuming four medium eggs per day for the duration of the study?

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn N Starr, PhD, RDN, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No